CLINICAL TRIAL: NCT07185321
Title: An Open-Label, Phase 1 Study to Investigate the Absolute Bioavailability and the Absorption, Metabolism, and Excretion of [14C]-Mosliciguat in Healthy, Adult Males
Brief Title: A Phase 1 Study of Mosliciguat in Healthy, Adult Males
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmovant, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: RVT-2301-106
Record Dates: First submitted 2025-09-12; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Dry Powder Inhalers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Mosliciguat (RVT-2301) (Experimental): Mosliciguat administered daily via dry powder inhaler.
  Interventions: Drug: Mosliciguat; Device: Dry Powder Inhaler
- 14C mosliciguat (Experimental): Administered orally and via IV
  Interventions: Drug: 14C mosliciguat

INTERVENTIONS:
Drug: Mosliciguat — Dose level for inhalation
  Arms: Mosliciguat (RVT-2301)
Drug: 14C mosliciguat — Dose level
  Arms: 14C mosliciguat
Device: Dry Powder Inhaler — Dry powder inhaler for mosliciguat
  Arms: Mosliciguat (RVT-2301)

SUMMARY:
This is a single-center, Phase 1, open-label, 3-period, fixed-sequence study to investigate the bioavailability, absorption, metabolism, excretion and the safety of mosliciguat administered to healthy male adults.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing and able to provide informed consent.
* Considered to be in good health by the Investigator, as determined by medical history, physical examination, vital sign measurements, 12 lead electrocardiogram (ECG), and laboratory test results.

Exclusion Criteria:

* History or presence of any condition (e.g., chronic diarrhea, urinary incontinence), or prior surgery (e.g., gastric bypass) that, in the opinion of the Investigator, poses a significant risk to participant safety and/or achievement of study objectives
* History or presence of COPD, moderate or persistent asthma, other chronic lung disease, or chronic respiratory condition within the last 5 years
* Acute or recent respiratory infection symptoms not resolved at least 3 days prior to Period 1 check-in.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Determine the absolute bioavailability (ABA) of mosliciguat following administration of a single inhaled dose of mosliciguat followed by an IV microtracer dose of [14C]-mosliciguat in healthy adult males | Baseline, Day 7
  Absolute bioavailability of inhaled mosliciguat
Area under the concentration-time curve (AUC) for mosliciguat | Baseline, Day 7
Assess the mass balance (i.e., cumulative excretion in urine and feces compared to the administered amount of radioactive isotope) of [14C] following a single oral dose of mosliciguat solution | Baseline, Day 28
  Urine and fecal recovery of total [14C] radioactivity, [14C]-mosliciguat
Maximum observed concentration (Cmax) | Baseline, Day 7

SECONDARY OUTCOMES:
Evaluate the incidence of Treatment-Emergent Adverse Events (safety and tolerability of mosliciguat) | Baseline, Day 44
  Incidence, nature, and severity of participant TEAEs, SAEs, and AEs

CONTACTS AND LOCATIONS:
Overall Officials: Ubaldo Martin, Study Director — Pulmovant, Inc.
Locations (1):
- Pharmaron, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No